The Impact of Standardized Tobacco Product Packaging on Young Adults in the Retail Environment NCT05973981 October 7, 2025

## **Study Protocol**

**Study objective.** The overall aim of this research is to experimentally evaluate the extent to which partially standardizing the color of tobacco packaging influences motivation to quit smoking cigarettes among young adults. The study took place in the RAND StoreLab, a life-sized replica of a convenience store.

**Study design.** The experimental conditions that we will compare in this study are: 1) Status Quo (Cigarette packages appear as they normally do - no standardization); 2) Partial standardization (Cigarette packages appear with half of the package using a standardized color); and 3) Full standardization (Cigarette packages appear with the entire package covered with a standardized color).

**Methods.** The study was approved by the RAND Human Subjects Protection Committee. Young adult cigarette smokers were recruited from the community through standard advertising campaigns. Interested individuals completed an internet screening to determine eligibility. Eligible individuals completed informed consent. Participants completed a baseline questionnaire that assessed demographics, and smoking and tobacco use. Participants were then randomized to one of the three experimental conditions. They were provided with a \$20 (fake) RSL gift card and asked to shop in the RSL for whatever they wanted, for as long as they wanted. They were asked to purchase at least one item and check-out and pay for the item(s) as they would in any convenience store. A confederate who was not involved in the consent or survey process served as the cashier. This cashier scanned the selected items for a total price, scanned the gift card, and bagged the items. After exiting the RSL, participants completed the main outcome measure, motivation to quit cigarettes. They then: underwent a graduated debriefing; were asked to guess the study's purpose; and were told that they would be unable to retain the items they selected from the RSL. Finally, they received compensation for participating.

**Statistical analysis plan.** First, we evaluated whether randomization distributed preshopping baseline characteristics evenly across the experimental conditions. These univariable analyses used either t-tests or chi-squared tests to evaluate significance (depending on variable distribution). Next, we used linear regression to evaluate the relationship between the experimental conditions and post-RSL shopping motivation to quit cigarettes. Models adjusted for age, gender, and race.